CLINICAL TRIAL: NCT01270230
Title: A Randomized Controlled Trial of the Bruthas Project
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01MH09089901-A1; R01MH090899 (NIH)
Record Dates: First submitted 2010-12-02; First posted 2011-01-05 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: HIV Infection
Keywords: HIV Prevention Intervention; African American Men who have Sex with Men
MeSH Terms: conditions — HIV Infections | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison Group, Standard HIV-CT (Experimental): The comparison group will receive standardized HIV counseling and testing (HIV-CT), with referrals to case management.
  Interventions: Behavioral: Standard HIV Testing and Counseling
- Intervention Group, Bruthas Counseling (Experimental): Participants assigned to this arm receive four individual HIV prevention counseling sessions.
  Interventions: Behavioral: Bruthas Project

INTERVENTIONS:
Behavioral: Bruthas Project — The Bruthas Project HIV prevention intervention is a four-session, semi-structured individual risk reduction counseling program based on the Information-Motivation-Behavior (IMB) theoretical model. The counseling sessions are designed to complement standardized HIV-Counseling and Testing, and are delivered every 2-3 weeks over the course of 3 months. Each session lasts for approximately one hour, and is facilitated by a trained African American male counselor. The counselors engage with participants using open-ended questions and a non-judgmental, conversational style designed to elicit feedback on an individual's current level of HIV-related risk. The counselor then provides information and strengthens the participant's prevention skills.
  Arms: Intervention Group, Bruthas Counseling
Behavioral: Standard HIV Testing and Counseling — This arm represents those receiving the standard HIV testing and counseling. We ultimately settled on the standard-of-care comparison group because our primary research question is whether the implementation of the intervention cast against the backdrop of usual care, in this case, HIV testing and counseling as mandated by the CDC, is efficacious. Thus, participants randomized to the comparison group will receive the current standard intervention which involves HIV testing, pre- and post-test counseling, plus linkage to case management. Individuals who test HIV-positive will be referred to post-test services including counseling for treatment options, HIV-positive support groups, and harm reduction workshops.
  Arms: Comparison Group, Standard HIV-CT

SUMMARY:
African American men who have sex with men and women (AAMSMW) are at particular risk for contracting and transmitting HIV, and represent a priority population for developing effective interventions. Despite the urgent need for effective prevention approaches for AAMSMW, to our knowledge no evidence-based HIV interventions have been developed and tested for this population. This study is a randomized controlled trial of the Bruthas Project(BP), an individual-level HIV prevention intervention, which builds on standardized HIV counseling and testing. Delivered in a series of four sessions by trained African American male counselors, the BP focuses on reviewing HIV transmission routes for male and female partners, strengthening sexual communication skills with both male and female partners, and improving condom use skills and other safer sex negotiation strategies. A randomized controlled trial of BP is necessary to determine the efficacy of the intervention and can lead to improved public health efforts at reducing HIV risk behavior among AAMSMW and in the African American community more generally. To evaluate the effect of the BP, the investigators will recruit and enroll a cohort of 400 AAMSMW who will be randomly assigned to either the intervention condition, in which they will be offered BP, or to the comparison condition, in which they will receive standardized HIV testing and counseling with referral to case management. The investigators will follow the cohort over 9 months and will assess participants at three time points: baseline, 3 months follow-up, and 6 months follow-up.

DETAILED DESCRIPTION:
African Americans account for half of all Americans currently living with AIDS, and men account for two-thirds of all African Americans with HIV. AAMSMW are at particular risk for contracting and transmitting HIV, and represent a priority population for developing effective interventions. Studies of AAMSMW conducted in multiple HIV-epicenters in the United States have reported high rates of unprotected intercourse with male and female partners, concurrent partnerships, and frequent substance use before sex, accompanied by non-disclosure and secrecy regarding sexual risk behaviors. These behavioral dynamics are likely to fuel transmission of HIV and other STDs in diverse sexual networks and communities. Despite the urgent need for effective prevention approaches for AAMSMW, to our knowledge no evidence-based HIV interventions have been developed and tested for this population.

We propose to test a behavioral prevention intervention, the BP, to reduce HIV-related sexual risk behavior among AAMSMW. The intervention was designed through four years of formative research with AAMSMW consisting of: (1) qualitative in-depth interviews, focus groups and field ethnography; (2) protocol and measure development; (3) pilot testing and evaluation; and (4) further refinement following process and preliminary outcome data. The BP counseling process was formulated on principles of the Information-Motivation-Behavior (IMB) theory of HIV prevention, and is characterized by an individual-level counseling process that is specifically tailored to recognize the social and cultural contexts that inform sexual behavior for AAMSMW. Delivered in a series of four sessions by trained African American male counselors, the BP focuses on reviewing HIV transmission routes for male and female partners, strengthening sexual communication skills with both male and female partners, and improving condom use skills and other safer sex negotiation strategies. Evidence thus far indicates that BP is an acceptable and feasible model for providing HIV prevention counseling to this population, and pilot outcome data show promising indications of behavior change. A team of trained BP staff have successfully utilized a multi-tiered outreach approach to identify AAMSMW, recruit eligible individuals, and engage and retain participants in a longitudinal evaluation design. A randomized controlled trial of BP is necessary to determine the efficacy of the intervention and can lead to improved public health efforts at reducing HIV risk behavior among AAMSMW and in the African American community more generally.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* African American
* Male
* History of sex with male and female partners in the past two years
* English speaker

Exclusion Criteria:

* participation in previous research with Bruthas Project
* non English speaker
* identifies as gay

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2011-02; Primary Completion 2015-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
sexual risk behavior with male and female partners | 9-months
  Our primary outcome measure will feature two approaches to assessing HIV risk: we will assess (a) general sexual risk behaviors during the past 3 months and (b) event-level characteristics of sexual risk episodes for the past 1 month. Participants will report on general sexual activity during the past 3 months, including insertive vaginal sex, insertive/receptive anal sex, and giving/receiving oral sex. They will report on overall number of episodes, number of unprotected episodes, and episodes by partner type (main, casual, paying) and by partner gender (male, female).

SECONDARY OUTCOMES:
HIV Testing | 9 months follow up
  We will ask participants the date of their most recent HIV test.

CONTACTS AND LOCATIONS:
Overall Officials: Emily A Arnold, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No